CLINICAL TRIAL: NCT01483287
Title: The Effects of Added Enzyme α-Galactosidase at a Carbohydrate-rich Meal in IBS
Brief Title: The Effects of Added Enzyme α-Galactosidase at a Carbohydrate-rich Meal in Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Simrén, Clinical Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nogasin
Record Dates: First submitted 2011-11-22; First posted 2011-12-01 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: Gastrointestinal Symptoms; Bloating; Distention
MeSH Terms: conditions — Irritable Bowel Syndrome; Dilatation, Pathologic | interventions — alpha-Galactosidase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Enzyme (Active Comparator): Capsules with alpha-galactosidase (enzyme) (400 GaIU x 3) are ingested at breakfast, lunch and dinner.
  Interventions: Dietary Supplement: Alpha-Galactosidase
- Placebo (Placebo Comparator): 3 capsules with a non-active substance are ingested at breakfast, lunch and dinner
  Interventions: Dietary Supplement: Alpha-Galactosidase

INTERVENTIONS:
Dietary Supplement: Alpha-Galactosidase — The study is conducted during a total of two days at two different occasions. Visit 1: The patients will be served breakfast and lunch at the gastro unit and dinner will be enclosed when the patient leave for home. At each meal (breakfast, lunch, and dinner) the participants will ingest three capsules with a total content of 1200 GaIU alpha-galactosidase-randomized to be either the enzyme (α-Galactosidase) or a non-active substance (placebo). Visit 2: The procedure from visit 1 will recur after at least two weeks has passed - except that the content of the capsules will be opposite from the first visit.
  No other food or beverage are ingested from 1800 hours the evening before the intervention day until breakfast the day after intervention (no exact time).
  Other Names: Nogasin

SUMMARY:
IBS (irritable bowel syndrome) is a functional gastrointestinal disorder which is characterized by recurrent pain and/or discomfort, altered stool form, and abdominal distension. It has been established that food items such as beans, peas, lentils, peppers, and onions can increase gas production. What these have in common is that they all contain large amounts of complex carbohydrates. The enzymes in the small intestine are not able to fully digest these large molecules, which in turn are fermented by the colonic microflora. This fermentation is conducted through the production of short chain fatty acids and gases such as hydrogen and methane. Alpha-Galactosidase is an enzyme that has the ability to break down these indigestible carbohydrates to galactose and sucrose in the small intestine and to facilitate the absorption and minimize the gas production from bacteria in the colon.

The aim of this study is to assess if the gastrointestinal symptoms, above all problems from gas and distension, is alleviated when the enzyme α-Galactosidase (present in Nogasin capsules) is ingested with food.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Irritable Bowel Syndrome(IBS), (in accordance with ROME III criteria), and
* With the specific symptoms of bloating and/or abdominal distension.

Exclusion Criteria:

* The patients should not have any other gastrointestinal diseases such as IBD or celiac disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in symptoms | 24 hours
  Symptom questionnaire are filled in each half hour during trial (hours 0800-1530),four times between hours 1700-2000, once at bedtime, once at following morning before breakfast. Changes between visit 1 and visit 2 are registered.

SECONDARY OUTCOMES:
Changes in expiration air | 24 hours
  The expiration air is analyzed each half hour between hours 0800-1530 to examine the content of methane and hydrogen gas. Changes between visit 1 and visit 2 are registered.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden